CLINICAL TRIAL: NCT04255862
Title: An Open-Label, Single-Center, Randomized, Parallel-Group, Single-Dose Bioequivalence Study of Bimekizumab Given as 1x2mL or 2x1mL Subcutaneous Injection in Healthy Study Participants
Brief Title: A Study to Evaluate the Bioequivalence of Bimekizumab Given as 1x2mL or 2x1mL Subcutaneous Injection in Healthy Study Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study recruitment temporarily halted due to difficulties executing the study under the COVID-19 pandemic
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0068; 2019-002378-30 (EudraCT Number)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy Study Participants
Keywords: UCB4940; Bimekizumab; Bioequivalence; Auto-injector; Healthy study participants; Safety-syringe
MeSH Terms: interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test 1 (Experimental): Study participants randomized to this arm will receive bimekizumab administered subcutaneously with bimekizumab-safety syringe-2 mL presentation (test 1).
  Interventions: Drug: Bimekizumab
- Reference 1 (Other): Study participants randomized to this arm will receive bimekizumab administered subcutaneously with a bimekizumab-safety syringe-1 mL presentation (reference 1).
  Interventions: Drug: Bimekizumab
- Test 2 (Experimental): Study participants randomized to this arm will receive bimekizumab administered subcutaneously with a bimekizumab-auto-injector-2 mL presentation (test 2).
  Interventions: Drug: Bimekizumab
- Reference 2 (Other): Study participants randomized to this arm will receive bimekizumab administered subcutaneously with a bimekizumab-auto-injector-1 mL (reference 2).
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Study participants will receive a single-dose of bimekizumab administered subcutaneously in the Treatment Period.
  Other Names: UCB4940; BKZ

SUMMARY:
The purpose of the study is to compare the pharmacokinetics (PK) of bimekizumab when administered subcutaneously (sc) as 1x2 mL versus 2x1 mL, using a bimekizumab-safety syringe presentation or bimekizumab-auto-injector presentation, in healthy study participants.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 years and ≤65 years of age inclusive, at the time of signing the informed consent
* Study participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory tests, during the Screening Visit and on admission
* Body weight minimum of 50 kg for male and 45 kg for female study participants and a maximum of 100 kg for all study participants, and body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive) at the Screening Visit

Exclusion Criteria:

* Study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Study participant has a known hypersensitivity to any excipients of bimekizumab (and/or an investigational device) as stated in this protocol
* Study participant has cardiovascular or cerebrovascular disease, including hypertension, angina, ischemic heart disease, transient ischemic attacks, stroke, peripheral arterial disease sufficient to cause symptoms, and/or requires therapy to maintain stable status
* Study participant has an active infection or history of infections as follows:

  1. Any active infection (except common cold) within 14 days prior to the Screening Visit
  2. A serious infection, defined as requiring hospitalization or iv anti-infectives within 2 months prior to the Screening Visit
  3. A history of opportunistic, recurrent, or chronic infections that, in the opinion of the Investigator, might cause this study to be detrimental to the study participant. Opportunistic infections are infections caused by uncommon pathogens (eg, pneumocystis jirovecii, cryptococcosis) or unusually severe infections caused by common pathogens (eg, cytomegalovirus, herpes zoster)
* Study participant has a history of a positive tuberculosis (TB) test or evidence of possible TB or latent TB infection at the Screening Visit
* Study participant has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection. Study participants who have evidence of, or tested positive for hepatitis B or hepatitis C are excluded
* Study participant has 12-lead ECG with changes considered to be clinically significant (eg, QT interval corrected using Fridericia's formula [QTcF] >450 ms, bundle branch block, or evidence of myocardial ischemia) at the Screening Visit or on Day -1
* Study participant has active neoplastic disease or history of neoplastic disease within 5 years of the Screening Visit (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care)
* Study participants receiving any live (includes attenuated) vaccination within the 8 weeks prior to the Screening Visit (eg, inactivated influenza and pneumococcal vaccines are allowed but nasal influenza vaccination is not permitted). Live vaccines are not allowed during the study or for 20 weeks after the dose of the investigational medicinal product (IMP)
* Study participant has previously participated in this study or the study participant has previously been assigned to treatment in a study of the medication under investigation in this study
* Study participant has participated in another study of an IMP (and/or an investigational device) within the previous 90 days or 5 half-lives, whichever is longer, prior to IMP administration
* Study participant has made a blood donation of a blood loss of more than 400 mL of blood or blood products within 90 days prior to admission (Day -1) or plans to donate blood during the study
* Study participant has a positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in real-time reverse transcriptase polymerase chain reaction (RT-PCR) on the admission sample
* Study participant has clinical signs and symptoms consistent with coronavirus disease 2019 (COVID-19), eg fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the previous 14 days prior to Screening or on admission
* Study participant who had severe course of COVID-19 (ie, hospitalization, extracorporal membrane oxygenation, mechanically ventilated)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0068 001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Data from Phase 1 trials in Healthy Volunteers is outside of UCB's data sharing policy and is unavailable for sharing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in February 2020 and concluded in April 2021.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS) which consisted of all randomized study participants.
Groups:
- Bimekizumab-SS-2mL (Test 1): Participants randomized to this arm received a single dose of bimekizumab 320 milligrams (mg) administered as a subcutaneous injection using a 2 milliliter (mL) safety syringe (SS) on Day 1 of the study.
- Bimekizumab-SS-2x1mL (Reference 1): Participants randomized to this arm received a single dose of bimekizumab 320 mg (2x160 mg) administered as a subcutaneous injection using 2x1 mL SS on Day 1 of the study.
- Bimekizumab-AI-2mL (Test 2): Participants randomized to this arm received a single dose of bimekizumab 320 mg administered as a subcutaneous injection using a 2 mL auto-injector (AI) on Day 1 of the study.
- Bimekizumab-AI-2x1mL (Reference 2): Participants randomized to this arm received a single dose of bimekizumab 320 mg (2x160 mg) administered as a subcutaneous injection using 2x1 mL AI on Day 1 of the study.
Period: Overall Study
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Started | 18 | 18 | 17 | 18
Completed | 18 | 18 | 17 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Full Analysis Set (FAS) which consisted of all randomized study participants who received full or partial investigational medicinal product (IMP) according to the treatment the study participants actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2) | Total
Number analyzed (Participants) | 18 | 18 | 17 | 18 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 16 | 16 | 66
  >=65 years | 1 | 1 | 1 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.8) | 51.1 (15.8) | 46.8 (15.7) | 46.7 (15.7) | 49.3 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 13 | 13 | 51
  Male | 6 | 5 | 4 | 5 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 17 | 17 | 18 | 69
  Other/Black | 0 | 1 | 0 | 0 | 1
  Other/Caucasian | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 18 | 18 | 17 | 18 | 71

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC) for a Single Dose Bimekizumab (BKZ)
Description: AUC is the area under the bimekizumab plasma concentration-time curve from time zero (Day 1 predose) to infinity.
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) was a subset of the FAS, consisting of those study participants who had no important protocol deviations affecting the PK variables and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*micrograms/milliliter (days*ug/mL)
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
days*micrograms/milliliter (days*ug/mL) | 1665 (34.2) | 1610 (31.3) | 1560 (19.1) | 1357 (35.5)
Statistical Analysis 1: Comparison: Bimekizumab-SS-2mL (Test 1) vs Bimekizumab-SS-2x1mL (Reference 1); Test type: Equivalence — Bioequivalence (BE) was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 80 to 125 for AUC; Geometric Mean Ratio = 103.4, 90% CI 2-sided [86.4 to 123.8]
Statistical Analysis 2: Comparison: Bimekizumab-AI-2mL (Test 2) vs Bimekizumab-AI-2x1mL (Reference 2); Test type: Equivalence — BE was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 80 to 125 for AUC; Geometric Mean Ratio = 115.0, 90% CI 2-sided [97.9 to 135.0]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) for a Single Dose Bimekizumab (BKZ)
Description: AUC0-t is the area under the bimekizumab plasma concentration-time curve from time zero (Day 1 predose) to the last observed quantifiable concentration.
Time Frame: From Baseline (Day 1 predose) at predefined time points to the last quantifiable concentration (Day 140)
Population: The PK-PPS was a subset of the FAS, consisting of those study participants who had no important protocol deviations affecting the PK variables and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*ug/mL
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
days*ug/mL | 1551 (31.4) | 1509 (29.2) | 1469 (17.5) | 1296 (33.7)
Statistical Analysis 1: Comparison: Bimekizumab-SS-2mL (Test 1) vs Bimekizumab-SS-2x1mL (Reference 1); Test type: Equivalence — BE was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 80 to 125 for AUC0-t; Geometric Mean Ratio = 102.8, 90% CI 2-sided [87.0 to 121.5]
Statistical Analysis 2: Comparison: Bimekizumab-AI-2mL (Test 2) vs Bimekizumab-AI-2x1mL (Reference 2); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 113.4, 90% CI 2-sided [97.4 to 131.9]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for a Single Dose Bimekizumab (BKZ)
Description: Cmax is the maximum observed plasma concentration.
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
ug/mL | 43.56 (26.8) | 41.90 (23.9) | 42.23 (20.3) | 36.94 (28.2)
Statistical Analysis 1: Comparison: Bimekizumab-SS-2mL (Test 1) vs Bimekizumab-SS-2x1mL (Reference 1); Test type: Equivalence — BE was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 80 to 125 for Cmax; Geometric Mean Ratio = 104.0, 90% CI 2-sided [90.3 to 119.7]
Statistical Analysis 2: Comparison: Bimekizumab-AI-2mL (Test 2) vs Bimekizumab-AI-2x1mL (Reference 2); Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 114.3, 90% CI 2-sided [99.5 to 131.4]

4. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE) From Baseline to End of Safety Follow-Up
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent adverse events (TEAEs) were defined as any event not present prior to the administration of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to study treatment.
Time Frame: From Baseline (Day 1) to end of Safety Follow-Up (up to Day 140)
Population: The FAS consisted of all randomized study participants who received full or partial IMP according to the treatment the study participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
percentage of participants | 66.7 | 44.4 | 70.6 | 38.9

5. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Serious Adverse Event (SAE) From Baseline to End of Safety Follow-Up
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose: a. Results in death, b. Is life-threatening, c. Requires inpatient hospitalization or prolongation of existing hospitalization, d. Results in persistent disability/incapacity, e. Is a congenital anomaly/ birth defect, f. Other important medical events which based on appropriate medical judgment, jeopardized the study participant and required medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline (Day 1) to end of Safety Follow-Up (up to Day 140)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
percentage of participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Description: Apparent terminal half-life, reported in units of days, as determined via simple linear regression (slope=-lambdaz) of natural log (ln) concentration versus time for data points in the terminal phase of the concentration-time curve. t1/2 is calculated as ln2/lambdaz.
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
days | 28.21 (17.3) | 27.24 (16.8) | 25.73 (27.8) | 22.84 (28.7)

7. Secondary Outcome: Time of Occurrence of the Maximum Observed Concentration (Tmax) of a Single Dose Bimekizumab (BKZ)
Description: tmax is the time to reach maximum plasma concentration.
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
Number analyzed (Participants) | 18 | 18 | 17 | 18
days | 6.981 [2.99 to 15.0] | 6.988 [2.92 to 12.0] | 6.943 [3.98 to 12.0] | 6.972 [3.00 to 8.98]

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) to end of Safety Follow-Up Visit (up to Day 140)
Description: Treatment-emergent adverse events (TEAEs) were defined as any event not present prior to the administration of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to study treatment. TEAEs were reported based on the Full Analysis Set.
Arm/Group | Bimekizumab-SS-2mL (Test 1) | Bimekizumab-SS-2x1mL (Reference 1) | Bimekizumab-AI-2mL (Test 2) | Bimekizumab-AI-2x1mL (Reference 2)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 12/18 | 8/18 | 12/17 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab-SS-2mL (Test 1) (N=18) | Bimekizumab-SS-2x1mL (Reference 1) (N=18) | Bimekizumab-AI-2mL (Test 2) (N=17) | Bimekizumab-AI-2x1mL (Reference 2) (N=18)
Eyelid haematoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema migrans (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 4 (4) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (8) | 4 (5) | 3 (5) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT04255862/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT04255862/SAP_001.pdf